CLINICAL TRIAL: NCT05218096
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Multicenter Study to Evaluate the Efficacy and Safety of ALXN2050 in Adult Participants With Generalized Myasthenia Gravis
Brief Title: Study of ALXN2050 in Adult Participants With Generalized Myasthenia Gravis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALXN2050-MG-201; 2021-001229-26 (EudraCT Number)
Record Dates: First submitted 2021-12-16; First posted 2022-02-01 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Generalized Myasthenia Gravis; Myasthenia Gravis
Keywords: ALXN2050; gMG
MeSH Terms: conditions — Myasthenia Gravis | interventions — rhoA GTP-Binding Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking of treatment allocation will be observed until at least Week 34.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ALXN2050: 180 mg (Experimental): Participants will receive ALXN2050.
  Interventions: Drug: ALXN2050
- ALXN2050: 120 mg (Experimental): Participants will receive ALXN2050.
  Interventions: Drug: ALXN2050
- Placebo (Placebo Comparator): Participants will receive placebo followed by ALXN2050.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALXN2050 — Oral tablet.
  Other Names: ACH-0145228 (formerly)
  Arms: ALXN2050: 120 mg; ALXN2050: 180 mg
Drug: Placebo — Oral tablet.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of ALXN2050 (120 milligrams [mg], 180 mg) in participants with generalized myasthenia gravis (gMG).

Safety will be monitored throughout the study.

DETAILED DESCRIPTION:
The study consists of a blinded 8-week Primary Evaluation Period (PEP) and a blinded 26-week Extended Treatment Period (ETP). After completion of 34 weeks of treatment, participants will enter an Open-label Extension (OLE) Period for up to 1.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MG at least 3 months (90 days) prior to the date of the Screening Visit. Confirmation of MG must be made via the following:

  1. Positive serologic test for anti AChR antibodies at the Screening Visit, and
  2. Abnormal neuromuscular transmission demonstrated by single fiber electromyography or repetitive nerve stimulation, or
  3. Positive response to an AChEI test (eg, edrophonium chloride test), or
  4. Improvement of signs or symptoms related to MG during treatment with an oral AChEI, as determined by the treating physician
* Myasthenia Gravis Foundation of America Clinical Classification Class II to IV at the Screening Visit.
* MG-ADL total score must be ≥ 5 (with at least 50% of the score attributed to non-ocular elements) at the Screening Visit and at randomization (Day 1).
* Participants receiving treatment with protocol-specified immunosuppressive therapies, corticosteroids, or acetylcholinesterase inhibitors must have been receiving treatment and on a stable dose prior to the date of the Screening Visit, with no changes to the regimen expected during screening, the PEP, and/or the ETP.

Exclusion Criteria:

* Estimated glomerular filtration rate ≤ 30 milliliters/minute/1.73 squared meters during Screening calculated by Chronic Kidney Disease Epidemiology Collaboration.
* History of thymectomy, thymomectomy, or any other thymic surgery within 12 months prior to the Screening Visit.
* Any untreated thymic malignancy, carcinoma, or thymoma. Participants with a history of treated thymic malignancy or carcinoma are eligible for enrollment if they meet pre-specified conditions outlined in the protocol.
* Clinical features consistent with Clinical Deterioration at the time of the Screening Visit or at any time during the Screening Period prior to randomization (Day 1).
* Use of the following within the time periods specified below:

  1. Intravenous immunoglobulin G or subcutaneous immunoglobulin within the 4 weeks (28 days) prior to the Screening Visit.
  2. Use of tacrolimus or cyclosporine within the 4 weeks (28 days) prior to the Screening Visit.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-04-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (17):
  - Research Site, Phoenix, Arizona
  - Research Site, Aurora, Colorado
  - Research Site, Boca Raton, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Tampa, Florida
  - Research Site, Lexington, Kentucky
  - Research Site, New Hyde Park, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, West Chester, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Springfield, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Milwaukee, Wisconsin
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
- Germany (5):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Düsseldorf
  - Research Site, Hamburg
  - Research Site, Leipzig
- Italy (7):
  - Research Site, Bergamo
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rome
  - Research Site, Udine
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Niš
- South Korea (3):
  - Research Site, Daegu
  - Research Site, Seoul
  - Research Site, Yangsan
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Seville
- Taiwan (3):
  - Research Site, Hualien City
  - Research Site, Taipei
  - Research Site, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN2050-MG-201&attachmentIdentifier=d7fb4ef2-75ad-45ff-9749-51566dbf9ca8&fileName=ALXN2050-MG-201_Abbreviated_CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study did not meet its primary efficacy endpoint and was early terminated by the Sponsor.
Groups:
- Group 1: ALXN2050 180 mg BID: Participants received 180 mg ALXN2050 BID during all 3 study periods (primary evaluation, extended treatment, open-label extension).
- Group 2: ALXN2050 120 mg BID: Participants received 120 mg ALXN2050 BID during all 3 study periods (primary evaluation, extended treatment, open-label extension).
- Group 3: Placebo: Participants received placebo BID during the primary evaluation period.
- Group 3a: Placebo/ALXN2050 180 mg BID: Participants received placebo BID during the primary evaluation period, followed by ALXN2050 180 mg BID during the extended treatment period and the open-label extension period.
- Group 3b: Placebo/ALXN2050 120 mg BID: Participants received placebo BID during the primary evaluation period, followed by ALXN2050 120 mg BID during the extended treatment period and the open-label extension period.
Period: Primary Evaluation
Arm/Group | Group 1: ALXN2050 180 mg BID | Group 2: ALXN2050 120 mg BID | Group 3: Placebo | Group 3a: Placebo/ALXN2050 180 mg BID | Group 3b: Placebo/ALXN2050 120 mg BID
Started | 28 | 14 | 28 | 0 | 0
Received at Least 1 Dose of Study Intervention (Full Analysis Set) | 28 | 14 | 28 | 0 | 0
Entered Extended Treatment Period | 27 | 14 | 26 | 0 | 0
Re-randomized to ALXN2050 120 mg BID | 0 | 0 | 13 | 0 | 0
Re-randomized to ALXN2050 180 mg BID | 0 | 0 | 13 | 0 | 0
Completed | 27 | 14 | 26 | 0 | 0
Not Completed | 1 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Period: Extended Treatment
Arm/Group | Group 1: ALXN2050 180 mg BID | Group 2: ALXN2050 120 mg BID | Group 3: Placebo | Group 3a: Placebo/ALXN2050 180 mg BID | Group 3b: Placebo/ALXN2050 120 mg BID
Started | 27 | 14 | 0 (All placebo participants completing the Primary Evaluation period were re-randomized to Group 3a and Group 3b.) | 13 (All Group 3 participants completing the Primary Evaluation period were re-randomized to Group 3a and Group 3b.) | 13 (All Group 3 participants completing the Primary Evaluation period were re-randomized to Group 3a and Group 3b.)
Received at Least 1 Dose of Study Intervention (Full Analysis Set) | 27 | 14 | 0 | 13 | 13
Entered Open-label Extension Period | 16 | 6 | 0 | 8 | 9
Completed | 16 | 6 | 0 | 8 | 9
Not Completed | 11 | 8 | 0 | 5 | 4
Not completed — Clinical Deterioration | 1 | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 6 | 3 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 2 | 2
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Period: Open-label Extension
Arm/Group | Group 1: ALXN2050 180 mg BID | Group 2: ALXN2050 120 mg BID | Group 3: Placebo | Group 3a: Placebo/ALXN2050 180 mg BID | Group 3b: Placebo/ALXN2050 120 mg BID
Started | 16 | 6 | 0 | 8 | 9
Received at Least 1 Dose of Study Intervention (Full Analysis Set) | 16 | 6 | 0 | 8 | 9
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 16 | 6 | 0 | 8 | 9
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 13 | 4 | 0 | 7 | 7

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all participants who received at least 1 dose of study intervention.
Groups:
- Group 3: Placebo/ALXN2050: Participants received placebo BID during the primary evaluation period, followed by re-randomization to Group 3a and Group 3b, after which they received ALXN2050 180 mg BID and ALXN205 120 mg BID, respectively, during the extended treatment period and open-label extension period.
- Total: Total of all reporting groups
Arm/Group | Group 1: ALXN2050 180 mg BID | Group 2: ALXN2050 120 mg BID | Group 3: Placebo/ALXN2050 | Total
Number analyzed (Participants) | 28 | 14 | 28 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (15.55) | 55.9 (13.02) | 58.2 (16.45) | 54.1 (15.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 10 | 38
  Male | 10 | 4 | 18 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — National Institutes of Health/Office of Management & Budget (NIH/OMB)
  Participants
    Hispanic or Latino | 4 | 1 | 1 | 6
    Not Hispanic or Latino | 24 | 13 | 26 | 63
    Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 4 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 26 | 10 | 27 | 63
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline MG-ADL Total Score [Mean (Standard Deviation); unit: units on a scale] — Myasthenia Gravis Activities of Daily Living (MG-ADL)
  units on a scale | 9.4 (2.23) | 9.0 (2.96) | 8.8 (1.75) | 9.1 (2.21)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Of Participants With a Myasthenia Gravis Activities of Daily Living (MG-ADL) Total Score Reduction Of ≥ 2 Points In Any 4 Consecutive Weeks During The First 8 Weeks And Who Did Not Receive Rescue Therapy
Description: The MG-ADL profile is an 8-item participant-reported scale that focuses on relevant symptoms and functional performance of ADL in participants with MG. The 8 items of the MG-ADL questionnaire were derived from symptom-based components of the original 13-item QMG scale to assess disability secondary to ocular (2 items), bulbar (3 items), respiratory (1 item), and gross motor or limb (2 items) impairment related to effects of MG. Each response is graded 0 (normal) to 3 (most severe). The MG-ADL total score was calculated as the sum of the scores of the 8 items and ranges from 0 to 24, with higher scores indicating worse function.
Time Frame: Baseline through Week 8
Population: Full Analysis Set: all participants who received at least 1 dose of study intervention. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Group 1: ALXN2050 180 mg BID: Participants received 180 mg ALXN2050 BID during the primary evaluation period.
- Group 2: ALXN2050 120 mg BID: Participants received 120 mg ALXN2050 BID during the primary evaluation period.
Arm/Group | Group 1: ALXN2050 180 mg BID | Group 2: ALXN2050 120 mg BID | Group 3: Placebo
Number analyzed (Participants) | 16 | 8 | 18
percentage of participants | 57.1 [40.0 to 73.1] | 57.1 [32.5 to 79.4] | 64.3 [47.0 to 79.2]
Statistical Analysis 1: Comparison: Group 1: ALXN2050 180 mg BID vs Group 3: Placebo; Test type: Other — Difference; p = 0.6797, Barnard's Unconditional Exact Test; Difference = -7.1, 90% CI 2-sided [-28.8 to 15.0] — CI calculated using the Chan and Zhang method
Statistical Analysis 2: Comparison: Group 2: ALXN2050 120 mg BID vs Group 3: Placebo; Test type: Other — Difference; p = 0.7341, Barnard's Unconditional Exact Test; Difference = -7.1, 90% CI 2-sided [-34.8 to 19.3] — CI calculated using the Chan and Zhang method

2. Secondary Outcome: Change From Baseline In Quantitative Myasthenia Gravis (QMG) Total Score At Week 8
Description: The QMG Score for Disease Severity is an objective evaluation of therapy for MG and is based on quantitative testing of sentinel muscle groups. The QMG instrument consists of 13 items: ocular (2 items), facial (1 item), bulbar (2 items), gross motor (6 items), axial (1 item), and respiratory (1 item); each graded 0 to 3, with 3 being the most severe. The QMG total score was calculated as the sum of the scores of the 13 items and ranges from 0 to 39, with higher scores indicating more severe disease. Baseline score at each timepoint as the response variable, treatment group, study visit, and treatment-by-study visit interaction as fixed categorical effects, and baseline QMG total score as a covariate were used to calculate the least square (LS) mean and the standard error.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group 1: ALXN2050 180 mg BID | Group 2: ALXN2050 120 mg BID | Group 3: Placebo
Number analyzed (Participants) | 28 | 13 | 27
units on a scale | -1.1 (0.67) | -3.0 (0.98) | -1.4 (0.68)

3. Secondary Outcome: Change From Baseline In MG-ADL Total Score At Week 8
Description: The MG-ADL profile is an 8-item participant-reported scale that focuses on relevant symptoms and functional performance of ADL in participants with MG. The 8 items of the MG-ADL questionnaire were derived from symptom-based components of the original 13-item QMG scale to assess disability secondary to ocular (2 items), bulbar (3 items), respiratory (1 item), and gross motor or limb (2 items) impairment related to effects of MG. Each response is graded 0 (normal) to 3 (most severe). The MG-ADL total score was calculated as the sum of the scores of the 8 items and ranges from 0 to 24, with higher scores indicating worse function. Baseline score at each timepoint as the response variable, treatment group, study visit, and treatment-by-study visit interaction as fixed categorical effects, and baseline MG-ADL total score as a covariate were used to calculate the LS mean and the standard error.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group 1: ALXN2050 180 mg BID | Group 2: ALXN2050 120 mg BID | Group 3: Placebo
Number analyzed (Participants) | 27 | 14 | 26
units on a scale | -2.5 (0.50) | -3.7 (0.70) | -3.2 (0.51)

4. Secondary Outcome: Change From Baseline In Quality Of Life In Neurological Disorders (Neuro-QoL) Fatigue Score At Week 8
Description: The Neuro-QoL Fatigue questionnaire is a reliable and validated brief 19-item survey of fatigue, completed by the participant. Each item is scored on a scale of 1-5, with 1 indicating "never" and 5 indicating "sometimes". The Neuro-QoL Fatigue score was calculated as the sum of the scores of the 19 items and ranges from 19-95, with higher scores indicating greater fatigue and greater impact of MG on activities. Baseline score at each timepoint as the response variable, treatment group, study visit, and treatment-by-study visit interaction as fixed categorical effects, and baseline Neuro-QoL Fatigue score as a covariate were used to calculate the LS mean and the standard error.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Group 1: ALXN2050 180 mg BID | Group 2: ALXN2050 120 mg BID | Group 3: Placebo
Number analyzed (Participants) | 28 | 13 | 27
units on a scale | -8.7 (2.65) | -10.1 (3.77) | -8.3 (2.73)

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to 30 days after last dose of study intervention (approximately 2 years).
Description: Safety Set: all randomized participants who received at least 1 dose of study intervention.
Groups:
- Group 1: ALXN2050 180 mg BID (Primary Evaluation): Participants received 180 mg ALXN2050 BID during the primary evaluation period.
- Group 2: ALXN2050 120 mg BID (Primary Evaluation): Participants received 120 mg ALXN2050 BID during the primary evaluation period.
- Group 3: Placebo (Primary Evaluation): Participants received placebo BID during the primary evaluation period.
- Group 1: ALXN2050 180 mg BID (Extended Treatment & Open-label Extension): Participants received 180 mg ALXN2050 BID during the extended treatment period and open-label extension period.
- Group 2: ALXN2050 120 mg BID (Extended Treatment & Open-label Extension): Participants received 120 mg ALXN2050 BID during the extended treatment period and open-label extension period.
- Group 3a: Placebo/ALXN2050 180 mg BID (Extended Treatment & Open-label Extension): Participants received placebo BID during the primary evaluation period, followed by ALXN2050 180 mg BID during the extended treatment period and the open-label extension period.
- Group 3b: Placebo/ALXN2050 120 mg BID (Extended Treatment & Open-label Extension): Participants received placebo BID during the primary evaluation period, followed by ALXN2050 120 mg BID during the extended treatment period and the open-label extension period.
Arm/Group | Group 1: ALXN2050 180 mg BID (Primary Evaluation) | Group 2: ALXN2050 120 mg BID (Primary Evaluation) | Group 3: Placebo (Primary Evaluation) | Group 1: ALXN2050 180 mg BID (Extended Treatment & Open-label Extension) | Group 2: ALXN2050 120 mg BID (Extended Treatment & Open-label Extension) | Group 3a: Placebo/ALXN2050 180 mg BID (Extended Treatment & Open-label Extension) | Group 3b: Placebo/ALXN2050 120 mg BID (Extended Treatment & Open-label Extension)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/14 | 0/28 | 0/27 | 0/14 | 1/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/28 | 1/14 | 3/28 | 4/27 | 4/14 | 3/13 | 2/13
Other Adverse Events (participants affected / at risk) | 17/28 | 7/14 | 15/28 | 17/27 | 7/14 | 9/13 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1: ALXN2050 180 mg BID (Primary Evaluation) (N=28) | Group 2: ALXN2050 120 mg BID (Primary Evaluation) (N=14) | Group 3: Placebo (Primary Evaluation) (N=28) | Group 1: ALXN2050 180 mg BID (Extended Treatment & Open-label Extension) (N=27) | Group 2: ALXN2050 120 mg BID (Extended Treatment & Open-label Extension) (N=14) | Group 3a: Placebo/ALXN2050 180 mg BID (Extended Treatment & Open-label Extension) (N=13) | Group 3b: Placebo/ALXN2050 120 mg BID (Extended Treatment & Open-label Extension) (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salmonella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0/18 (0) | 0/10 (0) | 0/10 (0) | 0/17 (0) | 0/10 (0) | 0/5 (0) | 1/4 (1) — Adverse event only affected female participants.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1: ALXN2050 180 mg BID (Primary Evaluation) (N=28) | Group 2: ALXN2050 120 mg BID (Primary Evaluation) (N=14) | Group 3: Placebo (Primary Evaluation) (N=28) | Group 1: ALXN2050 180 mg BID (Extended Treatment & Open-label Extension) (N=27) | Group 2: ALXN2050 120 mg BID (Extended Treatment & Open-label Extension) (N=14) | Group 3a: Placebo/ALXN2050 180 mg BID (Extended Treatment & Open-label Extension) (N=13) | Group 3b: Placebo/ALXN2050 120 mg BID (Extended Treatment & Open-label Extension) (N=13)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Macrocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid cyst (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 1 (1) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Demyelination (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (12) | 0 (0) | 5 (6) | 4 (5) | 1 (1) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ketonuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/10 (0) | 1/4 (1) | 0/18 (0) | 0/10 (0) | 0/4 (0) | 0/8 (0) | 0/9 (0) — Adverse events affected only male participants.
Cervical dysplasia (Reproductive system and breast disorders) | 0/18 (0) | 0/10 (0) | 0/10 (0) | 0/17 (0) | 0/10 (0) | 0/5 (0) | 1/4 (1) — Adverse events affected only female participants.
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spider vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study did not meet its primary efficacy endpoint and was early terminated by the Sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT05218096/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT05218096/SAP_001.pdf